CLINICAL TRIAL: NCT00083668
Title: A Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group, Dose-response Study to Evaluate the Efficacy and Safety of 3 Fixed Dosages of Paliperidone Extended Release (ER) Tablets and Olanzapine, With Open-label Extension, in the Treatment of Patients With Schizophrenia
Brief Title: Trial Evaluating Three Fixed Doses of Paliperidone Extended-Release (ER) Tablets and Olanzapine in the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004375
Record Dates: First submitted 2004-05-27; First posted 2004-05-28 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Olanzapine; PANSS; Extended release; Atypical neuroleptic
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The primary objective of the double-blind phase of this study is to evaluate the efficacy and safety of 3 fixed dosages of paliperidone ER (3, 9, and 15 mg/day) compared with placebo in adult patients with schizophrenia

DETAILED DESCRIPTION:
Paliperidone is being developed as a new therapeutic agent for the treatment of schizophrenia. The extended-release (ER) formulation of paliperidone was developed to deliver paliperidone at a relatively constant rate over a 24-hour period to improve the tolerability profile and decrease the potential for orthostatic hypotension. This study is designed to evaluate the efficacy and safety and tolerability of 3 dosages of paliperidone ER compared with placebo in adult patients with schizophrenia. This is a multicenter, double-blind, randomized, placebo- and active-controlled, parallel-group, dose-response study. Patients will be randomized into 1 of 5 treatment groups to receive oral dosages of paliperidone ER 3, 9, or 15 mg, olanzapine 10 mg, or placebo once daily for a 6-week period. The study includes a screening period of up to 5 days, followed by a 6-week double-blind treatment phase. Following the double-blind treatment phase, eligible patients (those who have completed the 6-week double-blind phase or who discontinue due to lack of efficacy after a minimum of 21 days) may enter the 52-week open-label extension with paliperidone ER monotherapy. While patients are hospitalized, efficacy will be assessed twice during the first week and at the end of the second week, and after patients are discharged from the hospital, they will return to have efficacy and safety assessments performed on a weekly basis through the end of the 6-week double-blind phase. Efficacy will be evaluated throughout the 6-week double-blind phase by completion of the Positive and Negative Syndrome Scale (PANSS), Clinical Global Impression Scale - Severity (CGI-S), Personal and Social Performance Scale (PSP), and Schizophrenia Quality of Life Scale, Revision 4 (SQLS-R4). The primary efficacy response will be measured by the change from baseline score to end of double-blind phase for PANSS total score. Safety will be monitored throughout the study and includes assessments of the incidence of adverse events; measurement of extrapyramidal symptoms using 3 rating scales (Abnormal Involuntary Movement Scale [AIMS], Barnes Akathisia Rating Scale [BARS], Simpson-Angus Rating Scale [SAS]); measurement of vital signs (laying down and standing blood pressure, pulse, temperature); electrocardiograms; and clinical laboratory tests. Double-blind phase: 3, 9, 15 mg of paliperidone ER, 10 mg of olanzapine or placebo taken orally once a day for 6 weeks.

Open-label phase: start on paliperidone ER 9 mg orally once a day; maintained on a flexible oral dosage of paliperidone ER (3, 6, 9, 12, or 15 mg/day) for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Double-blind phase: DSM-IV diagnosis of schizophrenia for at least 1 year
* experiencing an acute episode, with a total PANSS score at screening between 70 and 120
* agree to voluntary hospitalization for a minimum of 14 days
* willing and able to fill out self-administered questionnaires
* must be able to be compliant with self-administration of medication, or have consistent help/support available.

Open-label phase: have completed the 6 weeks of double-blind treatment or completed at least 21 days of treatment and discontinued due to lack of efficacy

* patient and investigator must agree that open-label treatment is in the best interest of the patient.

Exclusion Criteria:

* Double-blind phase: DSM-IV axis I diagnosis other than schizophrenia
* DSM-IV diagnosis of substance dependence within 6 months prior to screening evaluation (nicotine and caffeine dependence are not exclusionary)
* history of tardive dyskinesia or neuroleptic malignant syndrome (NMS)
* history of any severe preexisting gastrointestinal narrowing (pathologic or iatrogenic)
* previous history of a lack of response (2 adequate trials) to any antipsychotic
* significant risk of suicidal or violent behavior. Open-label extension: patients believed by the investigator to be at significant risk for suicidal or violent behavior
* received an injection of a depot antipsychotic since entry into the preceding double-blind phase.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2004-04; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total PANSS score to the end of the double-blind phase.

SECONDARY OUTCOMES:
Changes from baseline to the end of the double-blind phase in PSP, CGI-S, and SQLS-R4.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Davidson M, Emsley R, Kramer M, Ford L, Pan G, Lim P, Eerdekens M. Efficacy, safety and early response of paliperidone extended-release tablets (paliperidone ER): results of a 6-week, randomized, placebo-controlled study. Schizophr Res. 2007 Jul;93(1-3):117-30. doi: 10.1016/j.schres.2007.03.003. Epub 2007 Apr 26. PMID 17466492
- [Result] Meltzer HY, Bobo WV, Nuamah IF, Lane R, Hough D, Kramer M, Eerdekens M. Efficacy and tolerability of oral paliperidone extended-release tablets in the treatment of acute schizophrenia: pooled data from three 6-week, placebo-controlled studies. J Clin Psychiatry. 2008 May;69(5):817-29. doi: 10.4088/jcp.v69n0515. PMID 18466043
- See also: Trial Evaluating Three Fixed Doses of Paliperidone Extended-Release (ER) Tablets and Olanzapine in the Treatment of Patients With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=584&filename=CR004375_CSR.pdf